CLINICAL TRIAL: NCT02795819
Title: Phase 1 Study of the Pan-DAC Inhibitor AR-42 and Pazopanib in Advanced Soft Tissue Sarcoma and Renal Cell Carcinoma
Brief Title: Study of the Pan-DAC Inhibitor AR-42 and Pazopanib in Advanced Sarcoma and Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug no longer being clinically developed by manufacturer
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14-10774; NCI-2016-00851 (Registry Identifier: NCI CTRP); P30CA016059 (NIH)
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Renal Cell Carcinoma; Soft Tissue Sarcoma; Metastatic Disease
MeSH Terms: conditions — Carcinoma, Renal Cell; Sarcoma; Neoplasm Metastasis | interventions — HDAC-42; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort minus 1 (-1) (Experimental): Participants take 10 mg AR-42 orally per day on 3 non-consecutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 600mg orally daily continuously
  Interventions: Drug: AR-42; Drug: Pazopanib
- Cohort 1 (Experimental): Participants take 20 mg AR-42 orally per day on 3 non-consecutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 600mg orally daily continuously
  Interventions: Drug: AR-42; Drug: Pazopanib
- Cohort 2 (Experimental): Participants take 20 mg AR-42 orally per day on 3 non-consecutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 800mg orally daily continuously
  Interventions: Drug: AR-42; Drug: Pazopanib
- Cohort 3A (Experimental): Participants take 30 mg AR-42 orally per day on 3 non-consecutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 800mg orally daily continuously
  Interventions: Drug: AR-42; Drug: Pazopanib
- Cohort 3B (Experimental): Participants take 30 mg AR-42 orally per day on 3 non-consecutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 600mg orally daily continuously
  Interventions: Drug: AR-42; Drug: Pazopanib
- Cohort 4A (Experimental): Participants take 40 mg AR-42 orally per day on 3 non-consecutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 800mg orally daily continuously
  Interventions: Drug: AR-42; Drug: Pazopanib
- Cohort 4B (Experimental): Participants take 40 mg AR-42 orally per day on 3 non-consecutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 600mg orally daily continuously
  Interventions: Drug: AR-42; Drug: Pazopanib

INTERVENTIONS:
Drug: AR-42 — AR-42 tablets were taken orally once per day on 3 non-consecutive days during the first 3 weeks of each 4-week cycle. If treatment was interrupted during the cycle, the cycle was to be extended
  Other Names: HDAC-42; OSU-HDAC42
Drug: Pazopanib — Pazopanib tablets were taken orally once daily continuously during each 4-week treatment cycle. There were no scheduled breaks in pazopanib therapy
  Other Names: Votrient

SUMMARY:
This phase 1 study was developed to identify recommended phase 2 doses (RP2Ds) of AR-42 and pazopanib when given in combination for subsequent clinical trials and may have potentially identified candidate pharmacodynamic and predictive biomarkers.

DETAILED DESCRIPTION:
This study was a single-arm, open-label, dose escalation phase 1 trial to determine the RP2Ds of AR-42 and pazopanib when given in combination to patients with advanced Renal Cell Carcinoma (RCC) or Soft Tissue Sarcoma (STS). Eligible patients had recurrent, unresectable, or metastatic RCC or STS for which pazopanib was an appropriate therapy.

AR-42 was taken orally once per day on 3 non-consecutive days each week during the first 3 weeks of each 4-week cycle. Pazopanib was taken by mouth once daily continuously during each cycle.

A modified 3+3 dose-escalation design was to be followed until the maximum tolerated doses (MTDs) were determined. The initial cohort of patients were assigned to an AR-42 dose of 20 mg taken once per day on 3 non-consecutive days during the first 3 weeks of each 4-week cycle and a pazopanib dose of 600 mg once daily continuously. Additional patients would be enrolled until a total of 12 patients were treated at the MTDs.

The protocol specifies a dose escalation plan that initially impacts only the pazopanib dose. The starting dose of pazopanib (600 mg) was planned to be escalated early so that the FDA-approved full dose of pazopanib (800 mg) would be reached before escalating the AR-42 dose. In subsequent dose-escalation steps, the dose of AR-42 was planned to be increased in 10-mg increments from a starting dose of 20 mg to a maximum dose of 40 mg.

If the number of Dose-Limiting Toxicities (DLT) showed that the MTD was exceeded with a pazopanib dose of 800 mg , the pazopanib dose was planned to be decreased to 600 mg and the AR-42 dose increased in 10-mg increments regardless of relationship of the DLT to one or both study medications.

Toxicities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0). The DLT evaluation period was the first treatment cycle. A minimum of 6 doses of AR-42 and 21 doses of pazopanib were required for a patient to be DLT-evaluable (if DLT was not observed with the delivered dose). DLT was defined as any ≥ grade 3 toxicity occurring during the DLT evaluation period and attributed to one or both of the study medications EXCEPT the following:

* The first incidence of grade 3 PPE at any dose level (subsequent incidences of grade 3 PPE will be considered DLT)
* Grade 3 nausea and vomiting in the absence of adequate prophylaxis and/or responsive to medical management within 48 hours
* Grade 3 diarrhea in the absence of adequate prophylaxis and/or responsive to medical management within 48 hours
* Grade 3 fatigue responsive to medical management • Grade 3 asymptomatic hypertension lasting ≤ 7 days
* Grade 3 electrolyte abnormalities that are corrected within 48 hours and, when corrected, can be maintained
* Grade 3 asymptomatic lipase elevation lasting ≤ 7 days
* Grade 3 decrease in platelet count if no clinically significant hemorrhage has occurred
* Grades 3 and 4 decrease in white blood cell count
* Grade 3 decrease in neutrophil count
* Grade 4 decrease in neutrophil count lasting ≤ 7 days
* Grades 3 and 4 decrease in lymphocyte count

Dose escalation was planned to continue until the maximum-tolerated dose (MTD), defined as one dose level below the dose in which dose-limiting toxicities (DLTs) are observed in >1 of the participants (e.g., in at least 2 participants in a cohort of at least 3). In the cohort of 12 patients at the MTD, no more than 3 DLTs were allowed to confirm the MTD. The RP2D was defined as equal to or less than the MTD, with an allowance to consider an RP2D below the MTD given the overall tolerability of the regimen including the frequency of AEs that were not DLTs and the frequency of dose modifications.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent, unresectable, or metastatic Renal Cell Carcinoma (RCC) or Soft Tissue Sarcoma (STS) (any histologic type) for which pazopanib was an appropriate therapy
* Measurable or evaluable disease by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1200/mm3
  * Platelets ≥ 120,000/mm3
  * Hemoglobin ≥ 9.5 g/dL
* Adequate renal function as defined below:

  * Creatinine ≤ 1.5 x upper limit of normal (ULN) for the laboratory or calculated or actual creatinine clearance ≥ 60 mL/min
  * Proteinuria ≤ 2+ [100 mg/dL] (using a random urine sample or < 3.0 gm using a 24-hour sample) (Note: If urine sample indicates ≥ 2+ [100 mg/dL]), a 24-hour urine sample must be collected and tested; urine protein in the 24-hour sample must be < 3.0 gm/24 hours.)
* Adequate hepatic function as defined below:

  * Total bilirubin ≤ 1.5 x ULN for the laboratory (Note: Patients with known Gilbert's Syndrome were not eligible for this study)
  * Aspartate aminotransferase (AST) ≤ 2.5 x ULN for the laboratory
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN for the laboratory
* Non-hematologic toxicities from previous cancer therapies resolved to ≤ grade 1
* International normalized ratio (INR) ≤ 1.5
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN for the laboratory
* Left ventricular ejection fraction (LVEF) assessment (eg, echocardiogram, MUGA scan, first-pass technique) performed within 3 months prior to initiation of study treatment indicates an LVEF of ≥ 50%
* A woman of childbearing potential (WCBP), defined as a woman who was < 60 years of age and had not had a hysterectomy, must have had a documented negative serum pregnancy test within 7 days prior to initiating study treatment
* A WCBP and a male patient with a partner who was a WCBP must have agreed to use a medically accepted method for preventing pregnancy for the duration of study treatment and for 2 months following completion of study treatment
* Ability to have understood and willingness to have signed the consent form

Exclusion Criteria:

* Symptomatic or untreated brain metastasis
* Leptomeningeal metastasis
* Any investigational agent within 4 weeks prior to initiating study treatment
* Previous therapy with pazopanib
* Inability to swallow medication
* Known or suspected malabsorption condition or obstruction
* Contraindication to antiangiogenic agents, including:

  * Serious non-healing wound, non-healing ulcer, or bone fracture
  * Major surgical procedure or significant traumatic injury within 4 weeks prior to initiating study treatment; other surgical procedures within 2 weeks prior to initiating study treatment
  * Pulmonary hemorrhage/bleeding event ≥ grade 2 within 12 weeks prior to initiating study treatment
  * Any other hemorrhage/bleeding event ≥ grade 3 within 12 weeks prior to initiating study treatment
* History of organ allograft including corneal transplant
* Evidence of bleeding diathesis or coagulopathy
* Documented Gilbert's Syndrome
* Resting systolic blood pressure (BP) < 100 mmHg
* Hypertension defined as systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg despite optimal medical management
* QTc interval > 450 ms on screening 12-lead electrocardiogram (ECG)

  * If baseline QTc on screening ECG met exclusion criteria:

    * Check calcium, potassium, and magnesium serum levels.
    * Correct any identified hypocalcemia, hypokalemia, and/or hypomagnesemia and repeat ECG to reconfirm exclusion of patient due to prolonged QTc interval.
  * For patients with heart rate (HR) 60-100 bpm, manual read of QTc was not required.
  * For patients with a baseline HR < 60 bpm or > 100 bpm, manual read of the QT interval by a cardiologist was required, with Fridericia correction applied to determine QTc (ie, QTcF).
* Active or clinically significant cardiac disease including any of the following:

  * Unstable angina (eg, anginal symptoms at rest) or onset of angina within 3 months prior to initiating study treatment
  * Myocardial infarction within 6 months prior to initiating study treatment
  * Cardiac arrhythmias currently requiring anti-arrhythmic therapy other than beta blockers
* Any documented history of clinically significant thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident, transient ischemic attack, deep vein thrombosis, or pulmonary embolism necessitating therapeutic anticoagulation within 6 months prior to initiating study treatment (Note: Patients with a tumor-associated thrombus of locally-involved vessels were not excluded from participating in the study.)
* Active infection requiring treatment or chronic infection requiring suppressive therapy
* Chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Pleural effusion or ascites that caused respiratory compromise (eg, ≥ grade 2 dyspnea)
* Required ongoing treatment with other drugs thought to potentially have adverse interactions with either of the medications included in the study treatment; if such medications have been used, patients must have discontinued these agents at least 1 week prior to initiating study treatment. Examples include:

  * Strong CYP3A4 inhibitors and/or strong CYP3A4 inducers; the reference list of CYP isozymes and classification of strong, moderate, and weak interactions are available through the Food and Drug Administration (FDA website.
  * Strong inhibitors of P-glycoprotein (P-gp) and/or breast cancer resistance protein (BCRP); the reference list of strong inhibitors of P-gp and BCRP.
  * Simvastatin and other HMG-CoA reductase inhibitors (ie, statins)
  * Drugs that raise gastric pH including proton pump inhibitors and H2-blockers (Note: Short-acting antacids, in place of PPIs and H2-blockers, are permitted.)
  * HDAC inhibitors
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may have increased the patient's risk or limit the patient's adherence with study requirement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07-08; Primary Completion 2016-11-24 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a single academic medical center cancer clinic from July 8, 2016 through November 22, 2016.
Groups:
- Cohort 1: Participants take 20 mg AR-42 orally per day on 3 non-consectutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 600mg orally daily continuously
- Cohort 2: Participants take 20 mg AR-42 orally per day on 3 non-consectutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 800mg orally daily continuously
- Cohort 3A: Participants take 30 mg AR-42 orally per day on 3 non-consectutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 800mg orally daily continuously
- Cohort 3B: Participants take 30 mg AR-42 orally per day on 3 non-consectutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 600mg orally daily continuously
- Cohort 4A: Participants take 40 mg AR-42 orally per day on 3 non-consectutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 800mg orally daily continuously
- Cohort 4B: Participants take 40 mg AR-42 orally per day on 3 non-consectutive days during the 1st 3 weeks of each 4-week cycle and pazopanib 600mg orally daily continuously
Period: Overall Study
Arm/Group | Cohort Minus 1 (-1) | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B
Started | 0 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All baseline characteristics subjects were in Cohort 1
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 54.8 [38 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Recommended Phase 2 Doses (RP2Ds) of AR-42 and Pazopanib When Given in Combination.
Description: To determine the recommended phase 2 doses (RP2Ds) for AR-42 and pazopanib that are the same as or less than the maximum tolerated doses (MTDs). The dose-limiting toxicity (DLT) evaluation period will be the first treatment cycle. Patients must have taken a minimum of 6 AR-42 doses and a minimum of 21 pazopanib doses during cycle 1 to be considered evaluable for DLT, if DLT has not been observed at the delivered dose. Patients' treatment dose level, dose modification, evaluability for DLT, and DLTs will be listed and summarized by basic descriptive statistics such as frequency and proportion. The maximum tolerated dose(MTDs)/recommended phase 2 doses (RP2Ds) will be found based on the criteria in the protocol.
Time Frame: 1 month
Population: Incomplete objective. No maximum tolerated dose (MTD) nor recommended phase two dose (RP2D) identified. Two dose limiting toxicities observed in 6 patients treated at the first dose level. Study terminated prior to exploration of additional dose levels.
Measure: Count of Units; unit: Dose Limiting Toxicities
Units Other Than Participants: Dose Limiting Toxicities
Arm/Group | Cohort Minus 1 (-1) | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B
Number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0 | 0
Number analyzed (Dose Limiting Toxicities) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dose Limiting Toxicities | 0 | 2 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events That Were Related to Treatment, AR-42 and Pazopanib Combination.
Description: The safety and toxicity of AR-42 and pazopanib when given in combination. Adverse Events (AEs) were characterized and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0) to determine the safety and toxicity of the combination of AR-42 and pazopanib. All AEs regardless of grade were recorded from the beginning of the study procedures through 30 days following the end of study treatment.
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort Minus 1 (-1) | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B
Number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 6 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: The Antitumor Effects of the AR-42 and Pazopanib Treatment Regimen in Patients With Advanced Renal Cell Carcinoma (RCC) or Soft Tissue Sarcoma (STS).
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 5 months
Population: Of 6 patients treated at dose level 1, 4 were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort Minus 1 (-1) | Cohort 1 | Cohort 2 | Cohort 3A | Cohort 3B | Cohort 4A | Cohort 4B
Number analyzed (Participants) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Participants
  Partial Response | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Progression | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Cycle 1 Day 1 to Off-Study Visit for each patient. All trial patients were enrolled on Cohort 1.
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
General Disorders administration site conditions - Other, specify (General disorders) | 1 (2)
Multi Organ Failure (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Fibrinogen decreased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (6)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (8)
Bloating (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Malaise (General disorders) | 4 (9)
Non-cardiac chest pain (General disorders) | 1 (2)
Pain (General disorders) | 4 (5)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Blood bilirubin increased (Investigations) | 2 (4)
Creatinine increased (Investigations) | 2 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Investigations - Other, specify (Investigations) | 2 (3)
Lipase increased (Investigations) | 2 (5)
Lymphocyte count decreased (Investigations) | 6 (14)
Neutrophil count decreased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 4 (9)
Serum amylase increased (Investigations) | 1 (4)
Weight loss (Investigations) | 3 (4)
White blood cell decreased (Investigations) | 5 (10)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4)
Nausea (Metabolism and nutrition disorders) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 4 (4)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 3 (4)
Proteinuria (Renal and urinary disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Incomplete objectives due to early termination of trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT02795819/Prot_SAP_000.pdf